CLINICAL TRIAL: NCT06050473
Title: Preservation vs Sacrifice of the Supraclavicular Nerve During Clavicle ORIF: A Randomized Controlled Trial
Brief Title: Supraclavicular Nerve During Clavicle ORIF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: HealthPartners Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: A16-535
Record Dates: First submitted 2023-09-14; First posted 2023-09-22 (Actual); Last update posted 2023-09-22 (Actual); Status verified 2023-09

CONDITIONS: Clavicle Fracture
Keywords: Clavicle; Fracture; Supraclavicular nerve; Post-operative; Paresthesia
MeSH Terms: conditions — Fractures, Bone; Paresthesia

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants blinded to the cohort they are randomized to (i.e., nerve-sparing group vs nerve-sacrificing group). Care providers were blinded to the randomization and made aware of the patient's cohort just prior to surgery.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Supraclavicular nerve-sacrificing procedure (Active Comparator): Surgeon will not attempt to identify the supraclavicular nerve branches.
  Interventions: Procedure: Nerve-sacrificing procedure
- Supraclavicular nerve-preserving procedure (Active Comparator): Surgeon will attempt to dissect out, identify and preserve all branches of the supraclavicular nerve throughout the fracture reduction, fixation and closure.
  Interventions: Procedure: Nerve preserving procedure

INTERVENTIONS:
Procedure: Nerve-sacrificing procedure — Surgical fixation of the clavicle fracture will be performed through a horizontal incision over the clavicle. During the incision and soft tissue dissection, the surgeon will not attempt to identify the supraclavicular nerve branches. Instead, the surgeon will cut the nerve branches during the dissection.
  Arms: Supraclavicular nerve-sacrificing procedure
Procedure: Nerve preserving procedure — Surgical fixation of the clavicle fracture will be performed through the same horizontal incision over the clavicle. The surgeon will attempt to dissect out, identify and preserve all branches of the supraclavicular nerve throughout the fracture reduction, fixation and closure.
  Arms: Supraclavicular nerve-preserving procedure

SUMMARY:
Clavicle fractures are a common orthopedic injury and make up 2.6%-5% of all fractures. Despite the benefits of operative management, post-operative chest wall paresthesia is a well-known complication among surgeons and is well described in the literature. Studies reporting on the natural history of post-operative paresthesia report an incidence of chest wall numbness anywhere from 10-80% and this is attributed to iatrogenic injury of the branches of the supraclavicular nerve that provide sensation over the clavicle, anteromedial shoulder and proximal chest. While this may seem like an easy complication to avoid, anatomic studies give insight into the complex and unpredictable branching of the supraclavicular nerve. The aim of this study was to compare the area (cm2) and change in size over time of post-operative paresthesia (includes hypesthesia and dysesthesia) following ORIF of displaced clavicle fractures between nerve-sacrificing and nerve-preserving procedures.

DETAILED DESCRIPTION:
This is a prospective, partially-blinded, single center, randomized controlled trial to compare the post-operative outcomes of paresthesias and morbidity between nerve-preserving and nerve-sacrificing procedures after surgical fixation of clavicle fractures. Although prior studies explore different incision orientation, most fail to specify whether or not the supraclavicular nerve branches were identified and protected and also lack a patient questionnaire that focuses on paresthesia characteristics and patient quality of life as it relates to the measured area of postoperative numbness. In this proposed study, the investigators will be able to fill this gap in knowledge and give insight into whether or not a nerve-sparing technique should be used to decrease the morbidity of postoperative chest wall paresthesia following operative fixation of clavicle fractures. This research will be important to the scientific community because it will help guide a physician's pre-operative counseling and establish realistic expectations for their patients. It could also guide a physician's surgical technique in a manner to decrease post-operative morbidity for patient's undergoing surgical fixation of clavicle fractures.

1. Group 1 - Operative treatment utilizing a supraclavicular nerve-sacrificing procedure
2. Group 2 - Operative treatment utilizing a supraclavicular nerve-preserving procedure

ELIGIBILITY:
Inclusion Criteria:

* Patients >17 years old with a displaced, midshaft clavicle fracture
* Closed injury
* No skin compromise

Exclusion Criteria:

* Clavicle non-union/malunion
* Far proximal (medial) or far distal (lateral) clavicle fractures
* Open injury
* Skin compromise
* Prior surgery of the anterior chest wall or affected clavicle
* Pre-existing chest wall numbness, cervical root symptoms, neurologic or sensory deficits, signs of neuropathy
* We will not exclude patients on membrane stabilizing medications for nerve paresthesia (GABA agonists, tricyclic anti-depressants) but will include this on patient intake form and document it
* Traumatic brain injury
* Patients who had prior deltopectoral approach to glenoid

Min Age: 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2016-11-02 (Actual); Primary Completion 2023-08-10 (Actual); Study Completion 2023-08-10 (Actual)

PRIMARY OUTCOMES:
Paresthesia mapping | Each follow-up visit at 2 weeks post-operative, 12 weeks post-operative, 6 months post-operative, 1 year post-operative
  A trained research fellow will be blinded to the operative intervention performed and will measure the area of chest wall paresthesia using a transparency grid made up of 1cmx1cm squares. The transparency grid will be placed over the patient's clavicle and the patient will be instructed to palpate the chest wall for areas of paresthesia. The examiner will then outline the area of paresthesia by tracing it onto the transparency slide.

SECONDARY OUTCOMES:
Cutaneous Hyperesthesia/dysesthesia mapping | Each follow-up visit at 2 weeks post-operative, 12 weeks post-operative, 6 months post-operative, 1 year post-operative
  A 10 gram Semmes-Weinstein monofilament will be applied twice, for 1 second at each point as indicated on the diagram in Appendix E. It will be applied to two points at the medial 1/3, middle 1/3 and lateral 1/3 of the subclavicular region, 3cm distal the inferior border of the clavicle at each point. The monofilament will be applied twice for 1 second at each point. Unperceived points will be identified and recorded based on location at medial, middle or lateral 1/3. If this monofilament test results in dysesthesia (pain, tingling, shock like sensations), this will be recorded similarly.
Patient Morbidity | Prior to measuring the area of paresthesia each follow-up visit at 2 weeks post-operative, 12 weeks post-operative, 6 months post-operative, 1 year post-operative
  The research fellow will administer the Patient Morbidity questionnaire and record the patient's responses. This outlines the characteristics of the paresthesia and the effect on the patient. This will be the investigator's measure of patient-reported morbidity.
Disabilities of the Arm, Shoulder and Hand (DASH); A 30-item self-reported questionnaire in which the response options are presented as 5-point Likert scales. Scores range from 0 (no disability) to 100 (most severe disability). | Prior to measuring the area of paresthesia each follow-up visit at 2 weeks post-operative, 12 weeks post-operative, 6 months post-operative, 1 year post-operative
  The patient will fill out the Disability of Arm, Shoulder & Hand questionnaire as a measure of functional outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Peter A Cole, MD, Principal Investigator — HealthPartners Institute

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jeray KJ. Acute midshaft clavicular fracture. J Am Acad Orthop Surg. 2007 Apr;15(4):239-48. doi: 10.5435/00124635-200704000-00007. PMID 17426295
- [Background] Christensen TJ, Horwitz DS, Kubiak EN. Natural history of anterior chest wall numbness after plating of clavicle fractures: educating patients. J Orthop Trauma. 2014 Nov;28(11):642-7. doi: 10.1097/BOT.0000000000000095. PMID 24662990
- [Background] Ahrens PM, Garlick NI, Barber J, Tims EM; Clavicle Trial Collaborative Group. The Clavicle Trial: A Multicenter Randomized Controlled Trial Comparing Operative with Nonoperative Treatment of Displaced Midshaft Clavicle Fractures. J Bone Joint Surg Am. 2017 Aug 16;99(16):1345-1354. doi: 10.2106/JBJS.16.01112. PMID 28816894
- [Background] Canadian Orthopaedic Trauma Society. Nonoperative treatment compared with plate fixation of displaced midshaft clavicular fractures. A multicenter, randomized clinical trial. J Bone Joint Surg Am. 2007 Jan;89(1):1-10. doi: 10.2106/JBJS.F.00020. PMID 17200303
- [Background] Robinson CM, Goudie EB, Murray IR, Jenkins PJ, Ahktar MA, Read EO, Foster CJ, Clark K, Brooksbank AJ, Arthur A, Crowther MA, Packham I, Chesser TJ. Open reduction and plate fixation versus nonoperative treatment for displaced midshaft clavicular fractures: a multicenter, randomized, controlled trial. J Bone Joint Surg Am. 2013 Sep 4;95(17):1576-84. doi: 10.2106/JBJS.L.00307. PMID 24005198
- [Background] Ahmed AF, Salameh M, AlKhatib N, Elmhiregh A, Ahmed GO. Open Reduction and Internal Fixation Versus Nonsurgical Treatment in Displaced Midshaft Clavicle Fractures: A Meta-Analysis. J Orthop Trauma. 2018 Jul;32(7):e276-e283. doi: 10.1097/BOT.0000000000001174. PMID 29672340
- [Background] Nathe T, Tseng S, Yoo B. The anatomy of the supraclavicular nerve during surgical approach to the clavicular shaft. Clin Orthop Relat Res. 2011 Mar;469(3):890-4. doi: 10.1007/s11999-010-1608-x. Epub 2010 Oct 9. PMID 20936387
- [Background] Lemieux V, Afsharpour S, Nam D, Elmaraghy A. Incisional paresthesia following clavicle plate fixation: does it matter to patients? BMC Musculoskelet Disord. 2021 Nov 3;22(1):928. doi: 10.1186/s12891-021-04770-z. PMID 34732198
- [Background] Havet E, Duparc F, Tobenas-Dujardin AC, Muller JM, Freger P. Morphometric study of the shoulder and subclavicular innervation by the intermediate and lateral branches of supraclavicular nerves. Surg Radiol Anat. 2007 Dec;29(8):605-10. doi: 10.1007/s00276-007-0258-5. Epub 2007 Sep 13. PMID 17851634
- [Background] Jelev L, Surchev L. Study of variant anatomical structures (bony canals, fibrous bands, and muscles) in relation to potential supraclavicular nerve entrapment. Clin Anat. 2007 Apr;20(3):278-85. doi: 10.1002/ca.20368. PMID 16838268
- [Background] Wang K, Dowrick A, Choi J, Rahim R, Edwards E. Post-operative numbness and patient satisfaction following plate fixation of clavicular fractures. Injury. 2010 Oct;41(10):1002-5. doi: 10.1016/j.injury.2010.02.028. Epub 2010 Mar 12. PMID 20219192
- [Background] Erdogan M, Desteli EE, Imren Y, Kilic M, Ulusoy S, Varli A. Supraclavicular neuropathy after surgical treatment of clavicular fractures: comparison of two incisions. Acta Chir Orthop Traumatol Cech. 2014;81(6):387-91. PMID 25651293
- [Background] Chechik O, Batash R, Goldstein Y, Snir N, Amar E, Drexler M, Maman E, Dolkart O. Surgical approach for open reduction and internal fixation of clavicle fractures: a comparison of vertical and horizontal incisions. Int Orthop. 2019 Aug;43(8):1977-1982. doi: 10.1007/s00264-018-4139-9. Epub 2018 Sep 5. PMID 30187099
- [Background] Beirer M, Postl L, Cronlein M, Siebenlist S, Huber-Wagner S, Braun KF, Biberthaler P, Kirchhoff C. Does a minimal invasive approach reduce anterior chest wall numbness and postoperative pain in plate fixation of clavicle fractures? BMC Musculoskelet Disord. 2015 May 28;16:128. doi: 10.1186/s12891-015-0592-4. PMID 26018526
- [Background] Ko SH, Kim MS. Comparison of supraclavicular nerve injuries after clavicle mid-shaft surgery via minimally invasive plate osteosynthesis versus open reduction and internal fixation. Arch Orthop Trauma Surg. 2022 Aug;142(8):1895-1902. doi: 10.1007/s00402-021-03941-w. Epub 2021 May 9. PMID 33966101
- [Background] You JM, Wu YS, Wang Y. Comparison of post-operative numbness and patient satisfaction using minimally invasive plate osteosynthesis or open plating for acute displaced clavicular shaft fractures. Int J Surg. 2018 Aug;56:21-25. doi: 10.1016/j.ijsu.2018.06.007. Epub 2018 Jun 8. PMID 29890301
- [Background] Huang D, Deng Y, Cheng J, Bong YR, Schwass M, Policinski I. Comparison of patient reported outcomes following clavicle operative fixation using supraclavicular nerve sparing and supraclavicular nerve sacrificing techniques- A cohort study. Injury. 2021 Mar;52(3):501-505. doi: 10.1016/j.injury.2020.10.100. Epub 2020 Oct 27. PMID 33131791
- [Background] Meinberg EG, Agel J, Roberts CS, Karam MD, Kellam JF. Fracture and Dislocation Classification Compendium-2018. J Orthop Trauma. 2018 Jan;32 Suppl 1:S1-S170. doi: 10.1097/BOT.0000000000001063. No abstract available. PMID 29256945
- [Background] Laffosse JM, Potapov A, Malo M, Lavigne M, Vendittoli PA. Hypesthesia after anterolateral versus midline skin incision in TKA: a randomized study. Clin Orthop Relat Res. 2011 Nov;469(11):3154-63. doi: 10.1007/s11999-011-1973-0. Epub 2011 Jul 15. PMID 21761252
- [Background] O'Connor CM, Ring D. Correlation of Single Assessment Numeric Evaluation (SANE) with other Patient Reported Outcome Measures (PROMs). Arch Bone Jt Surg. 2019 Jul;7(4):303-306. PMID 31448305
- [Background] Amer K, Smith B, Thomson JE, Congiusta D, Reilly MC, Sirkin MS, Adams MR. Operative Versus Nonoperative Outcomes of Middle-Third Clavicle Fractures: A Systematic Review and Meta-Analysis. J Orthop Trauma. 2020 Jan;34(1):e6-e13. doi: 10.1097/BOT.0000000000001602. PMID 31851115
- [Background] Larsson S. Clavicula fractures: considerations when plating. Injury. 2018 Jun;49 Suppl 1:S24-S28. doi: 10.1016/S0020-1383(18)30298-5. PMID 29929688
- [Background] Devji T, Kleinlugtenbelt Y, Evaniew N, Ristevski B, Khoudigian S, Bhandari M. Operative versus nonoperative interventions for common fractures of the clavicle: a meta-analysis of randomized controlled trials. CMAJ Open. 2015 Nov 10;3(4):E396-405. doi: 10.9778/cmajo.20140130. eCollection 2015 Oct-Dec. PMID 26770963
- [Background] Ban I, Nowak J, Virtanen K, Troelsen A. Overtreatment of displaced midshaft clavicle fractures. Acta Orthop. 2016 Dec;87(6):541-545. doi: 10.1080/17453674.2016.1191275. Epub 2016 May 26. PMID 27225678
- [Background] O'Neill K, Stutz C, Duvernay M, Schoenecker J. Supraclavicular nerve entrapment and clavicular fracture. J Orthop Trauma. 2012 Jun;26(6):e63-5. doi: 10.1097/BOT.0b013e31822c0796. PMID 22430514